CLINICAL TRIAL: NCT03377348
Title: Evaluation of the Use of Intraoperative Subconjunctival Injection of Triamcinolone Acetonide and Limited Peritomy During Bare Scleral Pterygium Excision
Brief Title: Subconjunctival Injection of Triamcinolone Acetonide and Limited Peritomy During Pterygium Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Abdelhafez, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIP
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subconjunctival injection of triamcinolone acetonide (Other): intraoperative subconjunctival injection of triamcinolone acetonide and limited peritomy during bare scleral pterygium excision
  Interventions: Procedure: intraoperative subconjunctival injection of triamcinolone acetonide and limited peritomy during bare scleral pterygium excision

INTERVENTIONS:
Procedure: intraoperative subconjunctival injection of triamcinolone acetonide and limited peritomy during bare scleral pterygium excision — intraoperative subconjunctival injection of triamcinolone acetonide and limited peritomy during bare scleral pterygium excision

SUMMARY:
Pterygium is characterized by encroachment of a ﬂeshy fibrovascular tissue from the bulbar conjunctiva on to the cornea. Although previously thought to be a solely degenerative disease, a new evidence has demonstrated the role of cell proliferation and inflammation in the pathogenesis of pterygium , and also by the clinical data that steroids are beneﬁcial in halting progression of impending recurrent pterygium . Many techniques have been developed for pterygium surgery over time. The simple method of removing the head and body of pterygium and leaving the sclera uncovered, the so-called bare-sclera technique, has been associated with high recurrence rates of 32-88% . To reduce the recurrence rate after pterygium surgery with a bare-sclera technique, various adjunctive modalities have been used such as chemical agents including mitomycin C , 5-ﬂuorouracil . Furthermore, when removal of pterygium is accompanied with a graft, such as conjunctival autograft or amniotic membrane transplantation , lower recurrence rates have been achieved . However, it remains unclear why the bare sclera technique has poorer outcome with higher recurrence rate than other procedures.

DETAILED DESCRIPTION:
One of the factors that may have a role in the outcome of pterygium surgery is postoperative conjunctival inflammation , treatment of which has been demonstrated to improve the ﬁnal outcome . It has been shown that persistent conjunctival inflammation around the surgical site after pterygium surgery is present in 31-84% of cases with amniotic membrane transplantation, and in 15% of eyes with conjunctival autograft . However, the rate of conjunctival inflammation after pterygium surgery with a bare-sclera technique has not been reported in literature . Also, it has been suggested that higher recurrence rate after pterygium with amniotic membrane transplantation compared with conjunctival autograft may be due to higher rate of postoperative conjunctival inflammation . Therefore, it may be speculated that higher recurrence rate after pterygium surgery with a bare-sclera technique is partly due to higher rate of postoperative conjunctival inflammation .

ELIGIBILITY:
Inclusion Criteria:

* primary pterygium.

Exclusion Criteria:

* preexisting glaucoma .
* patient with family history of glaucoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
the rate of recurrence by grading system of Prabhasawat | 6 months
  it is a grade to follow up the recurrence of pterygium which classifies pterygium excision outcome from grades 1 to 4:
  * Grade 1 : indicates a normal appearance of the operated site .
  * Grade 2 : indicates the presence of fine episcleral vessels in the excised area, extending to the limbus but without any fibrous tissue .
  * Grade 3 : indicates fibrovascular tissue in the excised area, reaching to the limbus but not invading the cornea and significant conjunctival recurrence .
  * Grade 4: indicates a true corneal recurrence with fibrovascular tissue invading the cornea.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Abdelhafez, Master Degree, Principal Investigator — Assiut University
Locations (1):
- Alaa M. Abdelhafez, Asyut, Egypt